CLINICAL TRIAL: NCT06835829
Title: Comparing Advanced Hemostasis and Ultrasound-Guided Puncture to Conventional Approaches in Distal Radial Access: A Dual Randomized Pragmatic Trial
Brief Title: Comparing Advanced Hemostasis and Ultrasound-Guided Puncture to Conventional Approaches in Distal Radial Access
Acronym: ALPHA&OMEGA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associazione per lo Studio delle Malattie Cardiovascolari Cardiva ONLUS (Other)
Responsible Party: Principal Investigator, Gregory A. Sgueglia, Principal Investigator, S.Eugenio Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00123
Record Dates: First submitted 2025-02-01; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Coronary Catheterization
Keywords: Trasnradial access; Distal radial access; Ultrasound guidance; Potassium ferrate; Hemostasis

STUDY DESIGN:
Intervention Model Description: Prospective open-label, randomized, controlled trial that integrates two independent nonfactorial randomized comparisons.
  In the first comparison, 480 patients will be randomized in 1:1 ratio to either to conventional transradial access or distal radial access using the potassium ferrate patch for hemostasis enhancement.
  In the second comparison, the 240 patients assigned to distal radial access will be randomized 1:1 to either conventional artery puncture or ultrasound-guided puncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Distal radial access (Experimental)
  Interventions: Device: Distal radial potassium ferrate hemostatic patch
- Conventional transradial access (Active Comparator)
  Interventions: Device: Transradial potassium ferrate hemostatic patch
- Distal radial access ultrasound-guided (Experimental)
  Interventions: Procedure: Ultrasound-guidance
- Distal radial access conventional guidance (Active Comparator)
  Interventions: Procedure: Conventional guidance

INTERVENTIONS:
Device: Transradial potassium ferrate hemostatic patch — Use of a potassium ferrate hemostatic patch to enhance transradial access hemostasis
  Arms: Conventional transradial access
Device: Distal radial potassium ferrate hemostatic patch — Use of a potassium ferrate hemostatic patch to enhance distal radial access hemostasis
  Arms: Distal radial access
Procedure: Ultrasound-guidance — Ultrasound guidance for distal radial access
  Arms: Distal radial access ultrasound-guided
Procedure: Conventional guidance — Conventional guidance for distal radial access
  Arms: Distal radial access conventional guidance

SUMMARY:
Meta-analysis results show that distal radial access (DRA) is associated with a significant reduction in the risk of radial artery occlusion compared to conventional transradial access (TRA). This is of paramount importance in an evolving interventional context where an increasing number of radial access procedures are being performed to address a growing number of independent health conditions. DRA is also associated with a lower rate of vascular access-related adverse events, establishing it as the safest vascular access ever.

However, available data show that the success rate of DRA is lower than that of conventional TRA. Also, while the duration of hemostasis has been shown to be shorter, it has most likely not yet reached its full potential for shortening. Thus, the two extreme phases of DRA require important further evaluation.

The CompAring uLtrasound-guided Puncture and advanced HemostAsis to cOnventional approaches in distal radial access: a dual randoMizEd praGmatic triAl (ALPHA&OMEGA) trial will address this lack of knowledge by exploring whether a significantly shorter hemostasis duration can be achieved with DRA when using hemostasis enhancement and exploring whether ultrasound-guided puncture can increase the success rate of DRA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients presenting with CCS or ACS, including unstable angina or NSTEMI.
* Patients planned for coronary angiography or PCI.
* Patients able to provide written informed consent.
* Patient is willing to comply with all study protocol required evaluations.
* Palpable radial pulse both at conventional and distal puncture site.
* Reverse modified Barbeau test confirming radial artery patency in patients with a history of previous radial artery catheterization.

Exclusion Criteria:

* Acute ST-segment elevation myocardial infarction.
* Cardiogenic shock.
* Chronic hemodialysis.
* Contraindications to radial access, such as occlusive upper arm peripheral artery disease, or known anatomic variants prohibiting TRA on both sides.
* Medical conditions that may cause non-compliance with the study protocol and/or may confound the data interpretation.
* Patients unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Hemostasis duration. | From end of procedure to end of hemostasis (25 minutes for distal radial access and 60 minutes for conventional transradial access)
Access success | Starts when the anesthesia needle contacts the skin and stops when the introducer sheath has been properly placed (on average 1 minute)
  Access success occurs when an introducer sheath can be properly placed through the punctured artery.

IPD SHARING:
Plan to Share IPD: No